CLINICAL TRIAL: NCT01504243
Title: Association Between cd163 Gene Polymorphisms and Sepsis Among Chinese Han Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 20111013-009（1）; 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2012-01-04; First posted 2012-01-05 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-12

CONDITIONS: Sepsis
Keywords: CD163;; SNPs;; prognosis;; control（normal person）
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: normal person under medical examination
- sepsis: SIRS plus inflammation

SUMMARY:
CD163 is a member of the scavenger receptor cysteine-rich family (SRCR) is exclusively expressed on cells of the monocyte lineage.CD163 acts to amplify inflammation and serves as a critical mediator of inflammatory response in the context of sepsis. This study was designed to investigate whether CD163 genomic variations were associated with the prognosis of sepsis. We sequenced 30 sepsis patients with CD163 gene of seventeen exons by PCR sequencing. When analyzing the results of sequencing, we found five gene polymorphisms located in exon-2,exon-5 and exon-11, respectively. Compare with the NCBI dbSNP and Hapmap database, one polymorphisms located in exon-2 is non-synonymous variation rs3210140, two polymorphisms located in exon-5 are synonymous variations rs4883264 and rs4883263, the last two located in exon-11 are synonymous variations rs61729512 and rs150018775 . Five common polymorphisms (rs2234237,rs2234246) within the CD163 gene were detected in 200 patients with severe sepsis and in 200 healthy control subjects. This study was explored that whether or not polymorphisms detected within the CD163 gene may play a major role in the predisposition to prognosis of sepsis in a Chinese Han cohort.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis met the criteria recommended by 1991 ACCP/SCCM Joint Meeting and by the diagnostic criteria developed at the 2001 International Sepsis Definition Conference.

Exclusion Criteria:

* (1) younger than 18 years of age; (2) acquired immunodeficiency syndrome; (3) reduced polymorphonuclear granulocyte counts (< 500 μL-1); (4) died within 24h after admission into the ICU, or refused to participate in the study, or declined treatment during the period of observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between September 2009 and October 2011 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Li xin Xie, MD, Study Director — Respiratory Disease Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China